CLINICAL TRIAL: NCT07335458
Title: Free Play Surgery The Effects of Children's Fear and Anxiety and Parental Anxiety During the Intervention Process
Brief Title: Reducing Fear and Anxiety in Children Through Free Play
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Mustafa KARA, Principal Investigator, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E.229701
Record Dates: First submitted 2025-12-20; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Nursing
Keywords: Free play; Pediatric patient; Game-based intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental : Intervention group (Experimental): Children taken to the playground
  Interventions: Other: Entering the free play area
- Other: Game interference (No Intervention): Allowing patients in the intervention group to spend approximately 45 minutes in a free play area before surgery.

INTERVENTIONS:
Other: Entering the free play area — playing in the free play area before surgery
  Arms: Experimental : Intervention group

SUMMARY:
The aim of this study is to determine the effect of free play activities fear levels, and parental anxiety experienced before and after surgical intervention in children aged 4-10 years. The research is planned as a randomized controlled trial. The study population consists of children aged 4-10 years and their parents who will undergo planned surgical procedures in the pediatric surgery department of a university hospital. The sample will be selected using a convenience sampling method and will consist of individuals who volunteer to participate in the study. The data collection process in the study was planned in two stages, with experimental and control groups: pre-test and post-test. Tests for both groups will be administered prior to the planned surgical operation. A pre-test for the children and their parents in the experimental group will be administered approximately 2 hours before the surgical procedure, just before the start of the free play intervention. At this stage, baseline data will be obtained by measuring the children's fear and anxiety levels and the parents' anxiety levels. Following this, the children will be given approximately 30 minutes of free play. A post-test will be administered immediately after the play intervention, approximately 45 minutes before surgery. This measurement, along with the effect of free play on the dependent variables, will be used to evaluate the results. In the control group, no intervention will be applied, and routine procedures will continue. This group will also be assessed with a pre-test approximately 2 hours before surgery and a post-test approximately 30-60 minutes before surgery to evaluate their levels of fear and anxiety. This will allow for a comparison of any significant differences between the two groups. This timing aims to assess the children's anxiety and fear during the period when they experience the most intense anxiety and fear before surgery, and to validly measure the effectiveness of free play. Study Population: The study population consists of children aged 4-10 years who will undergo surgical intervention and their parents. Study Sample: The study will include children aged 4-10 years who require surgical intervention and their mothers and/or fathers. Participants will be randomly assigned to experimental and control groups. A review of similar studies in the literature shows that Sert (2023) worked with 70 people (35 experimental, 35 control group). Tuncay and Tüfekçi (2019) completed their research with 60 people, and Scarano et al. with 50 people. Similar to these studies, this study is planned to be completed with 70 people, 35 in the experimental group and 35 in the control group.

The hypotheses of the study are: H0.1: Free play has no significant effect on the fear and anxiety levels of children undergoing surgery. H1.1: The pre-operative fear and anxiety levels of children who underwent free play differ significantly from those in the control group. H0.2: Free play has no significant effect on the situational anxiety levels of parents whose children are undergoing surgery. H1.2: Free play has a significant effect on the situational anxiety levels of parents whose children are undergoing surgery. H0.3: There is no significant relationship between the mother's situational anxiety level and the child's fear and anxiety levels. H1.3: There is a significant relationship/difference between the mother's situational anxiety level and the child's fear and anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* The participant's age must be between 4-10 age range.
* The child's parent must agree to participate in the study voluntarily.

Exclusion Criteria:

* The participant's age must be outside the 4-10 age range.
* Having a chronic disease

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Children's State Anxiety Scale (CSA) score (0-10) | Baseline (preoperative, immediately before surgery)
  Children's State Anxiety (CSA) is a visual, thermometer-like self-report scale for children aged 4-10 years. The child is asked to mark how anxious/nervous they feel 'right now'. Scores range from 0 to 10. The child's mark is read using 0.5-point increments and then rounded to the nearest whole number; higher scores indicate greater state anxiety
Children's Fear Scale (CFS) score (0-4) | Baseline (preoperative, immediately before surgery)
  Children's Fear Scale (CFS) is a single-item faces scale consisting of five drawn facial expressions ranging from 0 (no anxiety/fear; neutral face) to 4 (severe anxiety/fear; frightened face). The scale will be completed independently by the child, the parent/caregiver, and a trained researcher. Scores range from 0 to 4; higher scores indicate greater fear/anxiety
Parental anxiety assessed by Visual Analog Scale (VAS, 0-100) | Baseline (preoperative, immediately before surgery)
  Parental anxiety is rated using a 0-100 mm Visual Analog Scale (VAS), where 0 indicates no anxiety and 100 indicates the worst imaginable anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa KARA, PhD, Principal Investigator — Osmaniye Korkut Ata University
Locations (1):
- Osmaniye Korkut Ata University, Osmaniye, Turkey (Türkiye)